CLINICAL TRIAL: NCT04014803
Title: Aspirin and a Potent P2Y12 Inhibitor Versus Aspirin and Clopidogrel Therapy in Patients Undergoing Elective Percutaneous Coronary Intervention for Complex Lesion Treatment (SMART-ATTEMPT)
Brief Title: Aspirin and a PoTent P2Y12 Inhibitor Versus Aspirin and Clopidogrel in Patients Undergoing PCI for Complex Lesion
Acronym: ATTEMPT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Inje University Ilsan Paik Hospital (Other); Seoul St. Mary's Hospital (Other); Mediplex Sejong Hospital (Unknown); Chonnam National University Hospital (Other); Sejong General Hospital (Other); Wonkwang University Hospital (Other); Gachon University Gil Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Chungbuk National University Hospital (Other); Yeungnam University Hospital (Other); Chungnam National University Hospital (Other); Wonju Severance Christian Hospital (Other); Konkuk University Chungju Hospital (Unknown); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Dankook University (Other); Incheon St.Mary's Hospital (Other); Gyeongsang National University Hospital (Other); Soonchunhyang University Hospital (Other); Ewha Womans University Seoul Hospital (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATTEMPT16453143
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Dual Antiplatelet Therapy; Complex Coronary Lesion
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prasugrel plus Aspirin arm (Active Comparator): Patients will receive 300 mg of aspirin before PCI unless they have previously received this antiplatelet medication. A loading dose of prasugrel 60 mg will be given before or after PCI as soon as possible following randomization, unless they have previously received the assigned medication. Aspirin 100 mg plus prasugrel 10 mg once daily* will be given for one year.
  * Based on previous studies including PRASFIT-ACS (PRASugrel compared with clopidogrel For Japanese patIenTs with ACS undergoing PCI) or TRILOGY ACS (The Targeted Platelet Inhibition to Clarify the Optimal Strategy to Medically Manage Acute Coronary Syndromes), maintenance dose can be reduced to 5 mg once daily in patients with high bleeding risk or by investigator's medical judgement.
  Interventions: Drug: Dual antiplatelet therapy with a P2Y12 inhibitor plus aspirin
- Clopidogrel plus Aspirin arm (Active Comparator): Patients will receive 300 mg of aspirin before PCI unless they have previously received this antiplatelet medication. A loading dose of clopidogrel 600 mg will be given before or after PCI as soon as possible following randomization, unless they have previously received the assigned medication. Aspirin 100 mg plus clopidogrel 75 mg once daily will be given for one year.
  Interventions: Drug: Dual antiplatelet therapy with a P2Y12 inhibitor plus aspirin

INTERVENTIONS:
Drug: Dual antiplatelet therapy with a P2Y12 inhibitor plus aspirin — Dual antiplatelet therapy with a P2Y12 inhibitor plus aspirin will be given according to the allocated arms in patients undergoing elective percutaneous coronary intervention for complex coronary lesion
  1. Prasugrel plus Aspirin arm
  2. Clopidogrel plus Aspirin arm
  Other Names: Prasugrel plus Aspirin or Clopidogrel plus Aspirin

SUMMARY:
This study is a prospective, open label, two-arm, randomized multicenter trial to evaluate the efficacy and safety of aspirin plus prasugrel as compared with aspirin plus clopidogrel in patients undergoing elective percutaneous coronary intervention with drug eluting stents for complex coronary lesions.

DETAILED DESCRIPTION:
Over the past several decades, dual antiplatelet therapy (DAPT) with the combination of aspirin and a P2Y12 inhibitor has become an essential treatment in patients undergoing percutaneous coronary intervention (PCI) to reduce ischemic events. Although the optimal duration of DAPT still remains controversial in patients with coronary artery disease, the recommended duration of maintenance of DAPT for patients undergoing PCI with drug-eluting stent is ≥12 months for those with acute coronary syndrome (ACS), and ≥6 months for those with stable coronary artery disease according to the current guidelines. However, individualized approach based on ischemic versus bleeding risks assessment is needed to determine the optimal duration of DAPT in various population.

Several studies reported that patients undergoing PCI for complex lesions had significantly higher rates of ischemic events than those with non-complex lesions. Moreover, prolonged DAPT of aspirin and clopidogrel more than 1 year significantly reduced the risk of cardiac ischemic events up to 44% in patients undergoing PCI for complex coronary lesions, and the current guideline recommends prolonged DAPT duration may be considered in patients undergoing complex PCI. Apart from prolonged use of DAPT, use of more potent P2Y12 inhibitor than clopidogrel may be another strategy to reduce ischemic events in patients undergoing PCI for complex coronary lesions. Prasugrel, a new thienopyridine, inhibits platelet aggregation more rapidly and potently than clopidogrel. In the TRITON-TIMI 38 (TRial to Assess Improvement in Therapeutic Outcomes by Optimizing Platelet InhibitioN with Prasugrel) study, prasugrel reduced ischemic events compared with clopidogrel in patients with acute coronary syndrome. Moreover, low dose prasugrel also reduced ischemic events without an excessive bleeding risk in Japanese population. Therefore, DAPT of aspirin and prasugrel would reduce recurrent ischemic events than DAPT of aspirin and clopidogrel in patients undergoing PCI for complex lesions, a high risk group of ischemic events, even when they do not present with myocardial infarction. So far, there have been no data on this issue.

The aim of the SMART-ATTEMPT (Aspirin and a PoTent P2Y12 inhibitor versus aspirin and clopidogrel Therapy in patients undergoing Elective percutaneous coronary intervention for coMPlex lesion Treatment) trial is to evaluate the efficacy and safety of aspirin plus prasugrel as compared with aspirin plus clopidogrel in patients undergoing elective PCI for complex lesions.

ELIGIBILITY:
Inclusion Criteria:

* ① Subject must be at least 19 years of age
* ② Subject who can verbally confirm understandings of risks, benefits and treatment alternatives and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure
* ③ Patients undergoing elective PCI as follows:

  1. True bifurcation lesion (Medina 1,1,1/1,0,1/0,1,1) with side branch ≥2.5 mm size
  2. Chronic total occlusion (≥3 months) as target lesion
  3. PCI for unprotected left main disease (left main ostium, body, or distal bifurcation including non-true bifurcation lesions)
  4. Long coronary lesions (expected stent length ≥38 mm)
  5. Multi-vessel PCI (≥2 vessels treated at one PCI session)
  6. Multiple stent needed (≥3 stents per patient)
  7. In-stent restenosis lesion as target lesion
  8. Severely calcified lesion (encircling calcium in angiography)
  9. Ostial lesions of left anterior descending artery, left circumflex artery, or right coronary artery

Exclusion Criteria:

* ① Hemodynamic instability or cardiogenic shock
* ② Subjects with serious bleeding (Intracerebral hemorrhage, gastrointestinal bleeding, hematuria, hemoptysis, and etc.)
* ③ Previous history of intracerebral hemorrhage, transient ischemic attack, or stroke
* ④ Known hypersensitivity or contraindications to study medications (aspirin, clopidogrel, and prasugrel)
* ⑤ Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
* ⑥ Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* ⑦ Patients presenting with biomarker positive acute coronary syndrome
* ⑧ Patients chronically taking prasugrel or ticagrelor (≥1 week)
* ⑨ Subjects ≥75 years of age or <60 kg of body weight
* ⑩ Patients taking warfarin or novel oral anticoagulants (dabigatran, rivaroxaban, edoxaban, or apixaban)

  * Eligible patients will be randomly assigned to treatment arms, stratified by participating centers, presence of diabetes mellitus, and stent types.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 1-year after randomization
  A composite of death, myocardial infarction, or stent thrombosis

SECONDARY OUTCOMES:
All-cause death | 1-year after randomization
  Death by any cause
Cardiac death | 1-year after randomization
  Death by cardiac cause
Myocardial infarction | 1-year after randomization
  Myocardial infarction
Stent thrombosis | 1-year after randomization
  Definite or probable stent thrombosis
Target lesion revascularization | 1-year after randomization
  Repeat revascularization for target lesion of index PCI
Target vessel revascularization | 1-year after randomization
  Repeat revascularization for target vessel of index PCI
Any revascularization | 1-year after randomization
  Any repeat revascularization
A composite of all-cause death/myocardial infarction/stent thrombosis/any revascularization | 1-year after randomization
  A composite of all-cause death/myocardial infarction/stent thrombosis/any revascularization
A composite of all-cause death/myocardial infarction | 1-year after randomization
  A composite of all-cause death/myocardial infarction
A composite of cardiac death/myocardial infarction | 1-year after randomization
  A composite of cardiac death/myocardial infarction
Cerebrovascular accident | 1-year after randomization
  Cerebrovascular accident
A composite of all-cause death/myocardial infarction/cerebrovascular accident | 1-year after randomization
  A composite of all-cause death/myocardial infarction/cerebrovascular accident
A composite of cardiac death/myocardial infarction/cerebrovascular accident | 1-year after randomization
  A composite of cardiac death/myocardial infarction/cerebrovascular accident
A composite of cardiac death/myocardial infarction/stent thrombosis | 1-year after randomization
  A composite of cardiac death/myocardial infarction/stent thrombosis
Bleeding by BARC types 3 or 5 | 1-year after randomization
  Bleeding defined by Bleeding Academic Research Consortium (BARC) types 3 or 5
Bleeding by BARC types 2, 3, or 5 | 1-year after randomization
  Bleeding defined by BARC types 2, 3 or 5
Net adverse clinical events | 1-year after randomization
  MACE + bleeding by BARC types 3 or 5

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea